CLINICAL TRIAL: NCT05248945
Title: Phase I, Open-Label, Single-Sequence Study of the Effect of Multiple Doses of Carbamazepine on Single-Dose Evobrutinib Pharmacokinetics in Healthy Participants
Brief Title: DDI Study of Evobrutinib and Carbamazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS200527_0108; 2021-003381-13 (EudraCT Number)
Record Dates: First submitted 2022-01-13; First posted 2022-02-21 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Clinical Pharmacology
MeSH Terms: interventions — evobrutinib; Carbamazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evobrutinib plus Carbamazepine (Experimental): Participants received a single oral dose of Evobrutinib 45 mg on Day 1 and Day 19 under fed condition followed by Cabamazepine 100 mg on Days 2 and 3, 200 mg on Days 4 and 5 and then 300 mg from Days 6 to 19 and were titrated back to 200 mg from Days 20 to 22 and 100 mg on Days 23 to 25 twice daily.
  Interventions: Drug: Evobrutinib; Drug: Carbamazepine

INTERVENTIONS:
Drug: Evobrutinib — Participants received a single oral dose of Evobrutinib 45 mg on Day 1 and Day 19
  Other Names: M2951
Drug: Carbamazepine — Participants received Carbamazepine 100 mg on Days 2 and 3, 200 mg on Days 4 and 5 and then 300 mg from Days 6 to 19 and were titrated back to 200 mg from Days 20 to 22 and 100 mg on Days 23 to 25 twice daily.

SUMMARY:
The purpose of this study was to investigate the effect of multiple doses of carbamazepine on two single doses of evobrutinib pharmacokinetics (PK) in healthy participants. Study details included:

Study Duration: up to 54 days. Treatment Duration: 25 days. Visit Frequency: Participants were residents in the Clinical Research Unit from Day 1 to Day 20 and returned on Day 26 for a Safety Follow-Up visit.

ELIGIBILITY:
Inclusion Criteria:

* Type of Participant and Disease Characteristics
* Had a body weight within 50.0 and 100.0 kg (kilogram) (inclusive) and Body Mass Index (BMI) within the range 19.0 and 30.0 kilogram per meter square (kg/m^2) (inclusive)
* Male: No contraception and barrier requirements were needed. Female: Was not a woman of childbearing potential
* Were capable of giving signed informed consent, which included compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and this protocol
* Were stable nonsmokers for at least 3 months preceding Screening

Exclusion Criteria:

* Had a history or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue, psychiatric (due to rare risk of hallucinations, agitation and activation of psychosis), and other diseases or disorders, and epilepsy, as determined by medical evaluation
* Had been administered live vaccines or live-attenuated virus vaccines within 3 months prior to Screening. Administration of other types of vaccines (e.g., SARSCoV2 vaccines) was allowed until 2 weeks before admission to Clinical Research Unit (CRU), thereafter it was prohibited until the end of the study
* Had been administered moderate or strong inhibitors or inducers of Cytochrome P450 (CYP)3A4/5 or Pgp within 4 weeks prior to the first administration of study intervention
* Had a contraindication to carbamazepine (carbamazepine SmPC)
* Had a history of any malignancy
* Had a history of drug hypersensitivity ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, including contact hypersensitivity to Electrocardiogram (ECG) electrodes, which may have affected the safety of the participant and/or outcome of the study per the Investigator's discretion.
* Other protocol defined exclusion criteria could have applied.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0108
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were planned out of which 14 participants received study drug.
Groups:
- Evobrutinib + Carbamazepine: Participants received a single oral dose of Evobrutinib 45 mg on Day 1 and Day 19 under fed condition followed by Cabamazepine 100 mg on Days 2 and 3, 200 mg on Days 4 and 5 and then 300 mg from Days 6 to 19 and were titrated back to 200 mg from Days 20 to 22 and 100 mg on Days 23 to 25 twice daily.
Period: Overall Study
Arm/Group | Evobrutinib + Carbamazepine
Started | 14
Completed | 12
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Elevated Gamma-Glutamyl Transferase (GGT) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero Extrapolated to Infinity (AUC0-inf) of Evobrutinib
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,16 and 24 hours post dose on Day 1 and Day 19.
Population: The Pharmacokinetic Analysis Set included all participants who had completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results. Here 'Overall number of participants analyzed' = number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter (h*ng/mL)
Groups:
- Evobrutinib: Participants received a single oral dose of Evobrutinib 45mg on Day 1.
- Evobrutinib + Carbamazepine: Participants received a single oral dose of Evobrutinib 45 milligram (mg) on Day 1 and Day 19 under fed condition followed by Cabamazepine 100 mg on Days 2 and 3, 200 mg on Days 4 and 5 and then 300 mg from Days 6 to 19 and were titrated back to 200 mg from Days 20 to 22 and 100 mg on Days 23 to 25 twice daily.
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 12
Hour*nanograms per milliliter (h*ng/mL) | 310 (33.2) | 49.2 (23.1)
Statistical Analysis 1: Comparison: Evobrutinib vs Evobrutinib + Carbamazepine; Test type: Other; Ratio of test and reference treatment = 15.83, 90% CI 2-sided [13.26 to 18.90]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Evobrutinib
Description: Cmax was obtained from plasma concentration time curve.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 16 and 24 hours post dose on Day 1 and Day 19.
Population: The Pharmacokinetic Analysis Set included all participants who had completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
nanogram per milliliter (ng/mL) | 132 (33.1) | 22.4 (33.1)
Statistical Analysis 1: Comparison: Evobrutinib vs Evobrutinib + Carbamazepine; Test type: Other; Ratio of test and reference treatment = 17.03, 90% CI 2-sided [13.59 to 21.33]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study intervention. A serious adverse event (SAE) was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE's were those events with onset dates on or after the first administration of study intervention. TEAEs include both Serious TEAEs and non-serious TEAEs."
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Participants
  Any TEAE | 14
  Any serious TEAE | 0

4. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, and Lymphocytes Values
Description: Blood samples were collected to analyze the hematology parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, and Lymphocytes Values. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
10^9 cells/Liter
  Platelets | 11 (34.0)
  Leukocytes | -0.23 (0.836)
  Neutrophils | -0.18 (0.857)
  Eosinophils | 0.04 (0.064)
  Basophils | 0.03 (0.027)
  Monocytes | -0.00 (0.111)
  Lymphocytes | -0.12 (0.541)

5. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Hemoglobin Levels
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin levels. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
grams per liter (g/L) | -5.178 (8.4346)

6. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Hematocrit Values
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit Value. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: litre of cells per litre of blood (L/L)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
litre of cells per litre of blood (L/L) | -0.014 (0.0236)

7. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Activated Partial Thromboplastin Time
Description: Blood samples were collected to analyze the hematology parameter: Activated Partial Thromboplastin Time. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
seconds | -0.6 (1.29)

8. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/ Leukocytes, and Neutrophils/Leukocytes
Description: Blood samples were collected to analyze the hematology parameter: basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/ leukocytes, and neutrophils/leukocytes. The data in terms of 'percentage of cells' was calculated as: Count of Basophils (10^9 cells/L) (or any other defined hematology parameter e.g. Neutrophils, Eosinophils etc.) divided by the total count of Leukocytes (10^9 cells/L) in the blood multiplied by 100."
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Percentage of cells
  Basophils/Leukocytes | 0.5 (0.44)
  Eosinophils/Leukocytes | 0.7 (0.98)
  Lymphocytes/Leukocytes | 0.1 (7.80)
  Monocytes/Leukocytes | 0.3 (2.11)
  Neutrophils/Leukocytes | -1.6 (8.95)

9. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Picograms | 0.35557 (0.506080)

10. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Femtoliter | 1.4 (0.93)

11. Secondary Outcome: Absolute Change From Baseline in Hematology Parameter: Prothrombin International Normalized Ratio
Description: Blood samples were collected to analyze the hematology parameter: Prothrombin International Normalized Ratio. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value. Percent=Fraction×100
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
percent | -0.04 (0.041)

12. Secondary Outcome: Absolute Change From Baseline in Biochemistry Parameter: Bilirubin, Creatinine and Urate
Description: Blood samples were collected to analyze the Biochemistry Parameter: Bilirubin, Creatinine and Urate. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: micromole/liter (umol/L)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
micromole/liter (umol/L)
  Bilirubin | -4.9 (2.91)
  Creatinine | -1 (8.2)
  Urate | -34.6 (59.35)

13. Secondary Outcome: Absolute Change From Baseline in Biochemistry Parameter: Sodium, Potassium, Calcium, Magnesium and Phosphate Levels
Description: Blood samples were collected to analyze the Biochemistry Parameter: Sodium, Potassium, Calcium, Magnesium and Phosphate Levels. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Millimoles per litre (mmol/L)
  Sodium Levels | 1 (1.6)
  Potassium Levels | 0.49 (0.407)
  Calcium Levels | 0.02 (0.084)
  Magnesium Levels | 0.05 (0.048)
  Phosphate Levels | 0.04 (0.210)

14. Secondary Outcome: Absolute Change From Baseline in Biochemistry Parameter: Protein and Albumin Levels
Description: Blood samples were collected to analyze the Biochemistry Parameter: Protein and Albumin Levels. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
g/L
  Protein | -4 (4.1)
  Albumin | 2.3 (2.61)

15. Secondary Outcome: Absolute Change From Baseline in Biochemistry Parameter: Alkaline Phosphatase, Amylase, Lipase, Creatinine Kinase, Gamma Glutamyl Transferase Levels, Lactate Dehydrogenase, Aspartate Aminotransferase
Description: Biochemistry Parameter: Alkaline Phosphatase, Amylase, Lipase, Creatinine Kinase, Gamma Glutamyl Transferase Levels, Lactate Dehydrogenase, Aspartate Aminotransferase. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Units per litre (U/L)
  Alkaline Phosphatase | 8 (11)
  Amylase | 1 (9.1)
  Lipase | 2 (3.48)
  Creatine Kinase | -33 (69.1)
  Gamma Glutamyl Transferase | 56 (49.4)
  Lactate Dehydrogenase | -1 (22.1)
  Aspartate Aminotransferase | 9 (14.3)

16. Secondary Outcome: Absolute Change From Baseline in Biochemistry Parameter: Glucose, Chloride, Cholesterol, Triglycerides, Phosphate Levels
Description: Biochemistry Parameter: Glucose, Chloride, Cholesterol, Triglycerides, Phosphate levels. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all subjects, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
mmol/L
  Glucose | 0.01 (0.439)
  Chloride | 2 (1.5)
  Cholesterol | 0.4 (0.60)
  Triglycerides | 0.2 (0.58)
  Phosphate | 0.04 (0.210)

17. Secondary Outcome: Absolute Change From Baseline in 12-Lead ECG Parameter: Heart Rate
Description: 12-Lead ECGs were collected after the participants rested quietly for at least 10 minutes in a supine position. 12-Lead ECG Parameter: Heart Rate. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
beats per minute | 2 (6.6)

18. Secondary Outcome: Absolute Change From Baseline in 12-Lead ECG Parameter: RR Duration, QT Duration, Fridericia's Formula (QTcF), PR Duration and QRS Duration
Description: 12-Lead ECGs were collected after the participants rested quietly for at least 10 minutes in a supine position. 12-Lead ECG Parameter: RR Duration. Baseline was the last scheduled measurement before administration of study intervention. Absolute changes from baseline were calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Millisecond (msec)
  RR Duration | -29 (94.9)
  QT Duration | -1 (8.7)
  QTcF | 2 (8.8)
  PR Duration | -2 (7.5)
  QRS Duration | -1 (3.9)

19. Secondary Outcome: Absolute Change From Baseline in Vital Sign: Blood Pressure
Description: Blood pressure (systolic and diastolic) was measured after at least 5 minutes resting, with the participant in the seated position without distractions.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Millimeters of mercury (mmHg)
  Systolic Blood Pressure | -2 (8.6)
  Diastolic Blood Pressure | -2 (4.8)

20. Secondary Outcome: Absolute Change From Baseline in Vital Sign: Pulse Rate
Description: Pulse rate was measured after at least 5 minutes resting, with the subject in the seated position without distractions.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per min
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
beats per min | 2 (7.3)

21. Secondary Outcome: Absolute Change From Baseline in Vital Sign: Respiratory Rate
Description: Respiratory Rate was measured after at least 5 minutes resting, with the participant in the seated position without distractions.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
breaths per minute | -1 (3.3)

22. Secondary Outcome: Absolute Change From Baseline in Vital Sign: Body Temperature
Description: The absolute changes from baseline in Body Temperature (degree Celsius [°C]) were reported.
Time Frame: Baseline Day 1 and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Degree Celsius | 0.1 (0.33)

23. Secondary Outcome: Total Body Clearance of Evobrutinib From Plasma (CL/f)
Description: CL/f was defined as the apparent total clearance of the drug from plasma after extravascular administration.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 12
Litres per hour (L/h) | 145 (33.2) | 914 (23.1)

24. Secondary Outcome: Apparent Volume of Distribution (Vz/f) of Evobrutinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. The apparent volume of distribution during the terminal phase following extravascular administration and was calculated by using the formula=Dose/ (AUC0-inf* λz).
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 12
Liter | 373 (20.0) | 1218 (28.4)

25. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-tlast) of Evobrutinib
Description: The AUC from time zero (= dosing time) to the time of the last quantifiable concentration (tlast).
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
h*ng/mL | 308 (33.4) | 46.1 (27.1)
Statistical Analysis 1: Comparison: Evobrutinib vs Evobrutinib + Carbamazepine; Test type: Other; Ratio of test and reference treatment = 14.98, 90% CI 2-sided [12.60 to 17.82]

26. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Evobrutinib
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
hours | 2.00 [0.500 to 4.00] | 2.00 [1.50 to 3.00]

27. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Evobrutinib in Plasma
Description: t1/2 was defined as the time taken for the plasma concentration or the amount of drug in the body to be reduced by half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 12
hours | 1.64 [0.997 to 2.89] | 0.961 [0.652 to 1.22]

28. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Evobrutinib Metabolite (MSC2729909A)
Description: as for outcome 1
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
hour*ng/mL | 115 (19.6) | 57.1 (20.1)
Statistical Analysis 1: Comparison: Evobrutinib vs Evobrutinib + Carbamazepine; Test type: Other; Ratio of test and reference treatment = 49.66, 90% CI 2-sided [44.93 to 54.90]

29. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (LOQ) (AUC0-tlast) of Evobrutinib Metabolite (MSC2729909A)
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration was at or above LOQ. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
h*ng/mL | 113 (19.7) | 55.7 (21.3)
Statistical Analysis 1: Comparison: Evobrutinib vs Evobrutinib + Carbamazepine; Test type: Other; Ratio of test and reference treatment = 49.41, 90% CI 2-sided [44.79 to 54.51]

30. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Evobrutinib Metabolite (MSC2729909A)
Description: Cmax was obtained from plasma concentration time curve.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
nanograms per milliliters (ng/mL) | 30.2 (23.4) | 21.0 (20.0)
Statistical Analysis 1: Comparison: Evobrutinib vs Evobrutinib + Carbamazepine; Test type: Other; Ratio of test and reference treatment = 69.65, 90% CI 2-sided [60.34 to 80.40]

31. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Evobrutinib Metabolite (MSC2729909A)
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
hours | 2.50 [0.500 to 4.0] | 2.50 [1.50 to 4.00]

32. Secondary Outcome: Time Prior to the First Quantifiable (Non-zero) Concentration (Tlag) of Evobrutinib Metabolite (MSC2729909A) in Plasma
Description: The time prior to the first concentration at or above limit of quantification. It is calculated as last time point at which the concentration is less than (<) Lower Limit of Quantification (LLOQ) before the occurrence of the first quantifiable concentration.
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
hours | 0.500 [0 to 1.52] | 0.500 [0 to 1.50]

33. Secondary Outcome: Metabolite to Parent Ratios for Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Evobrutinib Metabolite (MSC2729909A)
Description: Molecular weight-corrected ratio of metabolite (M) AUC0-inf to parent (P) AUC0-inf: M/P(AUC0-inf) = (AUC0-inf metabolite (MSC2729909A) *molecular weight (MW) parent) / (AUC0-inf parent*MW metabolite (MSC2729909A)).
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 12
Ratio | 0.344 (31.0) | 1.11 (21.7)

34. Secondary Outcome: Metabolite to Parent Ratios for Maximum Observed Plasma Concentration (Cmax) of Evobrutinib Metabolite (MSC2729909A)
Description: Molecular weight-corrected ratio of metabolite Cmax to parent Cmax: M/P(Cmax) = (Cmaxmetabolite (MSC2729909A) * MWparent) / (Cmax parent * MW metabolite (MSC2729909A)).
Time Frame: Evobrutinib: Predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,16 and 24 hours post dose on Day 1 and Day 19.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Evobrutinib | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 13 | 13
Ratio | 0.213 (23.6) | 0.870 (20.9)

35. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on Severity
Description: AE was defined as any untoward medical occurrence in a subject. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study intervention. SAE was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE's were those events with onset dates on or after the first administration of study intervention. TEAEs include both Serious TEAEs and non-serious TEAEs. Severity of AE were assessed by the investigator as Mild, Moderate, and Severe: An event that prevents normal everyday activities. Severe is a category used to rate the intensity of an event; both AEs and SAEs can be assessed as severe. SAS is used.
Time Frame: Baseline (Day 1) and Day 26
Population: The safety analysis set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib + Carbamazepine
Number analyzed (Participants) | 14
Participants
  Mild | 14
  Moderate | 7
  Severe | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Day 26
Arm/Group | Evobrutinib + Carbamazepine
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evobrutinib + Carbamazepine (N=14)
Diplopia (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Faeces hard (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Fatigue (General disorders) | 3
Feeling drunk (General disorders) | 1
Malaise (General disorders) | 1
Rash pustular (Infections and infestations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Aphasia (Nervous system disorders) | 1
Coordination abnormal (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 7
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 7
Agitation (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Listless (Psychiatric disorders) | 1
Terminal insomnia (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT05248945/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT05248945/SAP_001.pdf